CLINICAL TRIAL: NCT00916344
Title: Master Study of the EVIA DR-T/DR/SR-T/SR Pacemaker
Brief Title: Master Study for the Investigation of Safety and Efficacy of the EVIA Pacemaker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38-1
Record Dates: First submitted 2009-06-04; First posted 2009-06-09 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Pacemaker Indication

ARMS (1):
- Pacemaker therapy (Experimental)
  Interventions: Device: EVIA Pacemaker

INTERVENTIONS:
Device: EVIA Pacemaker — patient has standard indication for pacemaker therapy

SUMMARY:
The objective of this study is to prove the safety and efficacy of the EVIA pacemaker. Primarily, the newly implemented Atrial Capture Control algorithm is evaluated, which automatically measures the right atrial threshold and subsequently adjusts the pacing output.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for pacemaker therapy
* Understand the nature of the procedure
* Give informed consent
* Able to complete all testing required by the clinical protocol
* Available for follow-up visits on a regular basis at the investigational site

Exclusion Criteria:

* Meet none of the pacemaker indications
* Meet one or more of the contraindications
* Patients with chronic atrial fibrillation (dual chamber pacemaker only)
* Have a life expectancy of less than six months
* Cardiac surgery in the next six months
* Enrolled in another cardiac clinical investigation
* Have other medical devices that may interact with the implanted pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ritter, Dr., Principal Investigator — CHU Bordeaux Haut-Lévêque
Locations (1):
- CHU Bordeaux Haut-Lévêque, Pessac, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study the data of n = 175 patients from 34 clinical sites in Austria, Denmark, France, Germany, Spain, Sweden and United Kingdom are included. The period of investigation covered was between June 04, 2009 (day of first implant) and February 26, 2010 (day of last follow-up).
Groups:
- Pacemaker Therapy: Evia DR-T/ DR / SR-T / SR Single (SR) and dual (DR) chamber pacemaker with telemetry function (T)
Period: Overall Study
Arm/Group | Pacemaker Therapy
Started | 175
Completed | 167
Not Completed | 8
Not completed — Death | 2
Not completed — ICD upgrade | 1
Not completed — Drop-out | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 175
Age Continuous [Mean (Standard Deviation); unit: years] | 74 (10.5)
Age, Customized [Number; unit: participants]
  Between 34 and 93 years | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 92
Region of Enrollment [Number; unit: participants]
  Austria | 32
  Denmark | 19
  France | 9
  Germany | 93
  Spain | 16
  Sweden | 4
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Atrial Capture Control Feature (Automatic Atrial Threshold Test Minus Manual Atrial Measurement)
Description: atrial capture control: feature that automatically measures the atrial pacing threshold and subsequently adjusts the atrial pulse amplitude.
  atrial threshold test: measurable automatically or manually.
Time Frame: 1 month follow-up completed
Population: At 1 month follow-up 93 patients with dual chamber pacemaker had both manual and automatic atrial treshold tests (ITT analysis).
Measure: Mean (95% Confidence Interval); unit: Volt
Units Other Than Participants: (dual chamber pacemakers only at 1 mFU)
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 93
Number analyzed ((dual chamber pacemakers only at 1 mFU)) | 93
Volt | -0.01 [-0.03 to 0.02]

2. Secondary Outcome: Complication Free Rate
Description: Complication free rate (in %):
  1 minus(the number of possibly pacemaker related complications divided by the number of patients)
Time Frame: 1- and 3- month follow-up completed
Measure: Number (95% Confidence Interval); unit: Percentage complication free patients
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 175
Percentage complication free patients | 99 [96 to 100]

ADVERSE EVENTS:
Arm/Group | Pacemaker Therapy
Serious Adverse Events (participants affected / at risk) | 52/175
Other Adverse Events (participants affected / at risk) | 28/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=175)
Atrial fibrillation / flutter related (Cardiac disorders) | 3 (3)
ablation (Surgical and medical procedures) | 1 (1)
acute circulation insufficiency (Blood and lymphatic system disorders) | 1 (1)
bypass operation (Surgical and medical procedures) | 2 (2)
cardiac decompensation (Cardiac disorders) | 5 (7)
cardiogenic shock during implantation (Surgical and medical procedures) | 1 (1)
chest pain (Cardiac disorders) | 3 (3)
coronary angiography (Surgical and medical procedures) | 3 (3)
coronary artery disease related (Cardiac disorders) | 2 (2)
cystitis (Renal and urinary disorders) | 1 (1)
dementia (Nervous system disorders) | 1 (1)
diabetes related (Endocrine disorders) | 1 (3)
dialysis related (Renal and urinary disorders) | 1 (1)
fever and infection (Infections and infestations) | 1 (1)
foot amputation due to endocrine disorder (Surgical and medical procedures) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
intestinal disease (Gastrointestinal disorders) | 3 (3)
joint and bone related (Musculoskeletal and connective tissue disorders) | 2 (2)
lead dislocation (Surgical and medical procedures) | 10 (11)
lifestyle modification (Social circumstances) | 1 (1)
lung related hospitalisation (Respiratory, thoracic and mediastinal disorders) | 3 (3)
malnutrition (Metabolism and nutrition disorders) | 1 (1)
minor myocardial infarction (Cardiac disorders) | 1 (1)
noise hypersensibility (General disorders) | 1 (1)
non-cardiac death (Gastrointestinal disorders) | 1 (1)
non-cardiac death (Nervous system disorders) | 1 (1)
pacemaker/ICD exchange/repositioning (Surgical and medical procedures) | 3 (3)
pericardial effusion and pericardectomy (Surgical and medical procedures) | 1 (1)
pocket haematoma (Skin and subcutaneous tissue disorders) | 4 (4)
spinal disease (Nervous system disorders) | 4 (4)
stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=175)
Others (General disorders) | 11 (11)
circulation problems (Cardiac disorders) | 2 (2)
gastrointestinal disease (Gastrointestinal disorders) | 3 (3)
lead dislocation (Surgical and medical procedures) | 2 (2)
pacemaker related (Cardiac disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No